CLINICAL TRIAL: NCT00864812
Title: A Randomized, Open Label, Multicenter, Phase 4 Study for the Comparison of Efficacy of Tiotropium Plus Salmeterol/ Fluticasone Propionate Compared With Tiotropium Alone in COPD Patients
Brief Title: Clinical Outcomes of Tiotropium Plus Fluticasone Propionate/Salmeterol Compared With Tiotropium for Chronic Obstructive Pulmonary Disease (COPD) in Korea
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: The Korean Academy of Tuberculosis and Respiratory Diseases (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sung-Koo, Han /Chairman, The Korean Academy of Tuberculosis and Respiratory Diseases
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 112942
Record Dates: First submitted 2009-03-17; First posted 2009-03-19 (Estimated); Last update posted 2010-03-31 (Estimated); Status verified 2010-03

CONDITIONS: Chronic Obstructive Pulmonary Disease
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Tiotropium Bromide; Fluticasone; Salmeterol Xinafoate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): tiotropium with fluticasone propionate/salmeterol (FSC)
  Interventions: Drug: tiotropium with fluticasone propionate/salmeterol (FSC)
- 2 (Active Comparator): tiotropium
  Interventions: Drug: tiotropium

INTERVENTIONS:
Drug: tiotropium with fluticasone propionate/salmeterol (FSC) — COPD patients treated with tiotropium with fluticasone propionate/salmeterol (FSC)
  Other Names: tiotropium]:Spiriva; fluticasone propionate/salmeterol (FSC): Seretide
  Arms: 1
Drug: tiotropium — COPD patients treated with tiotropium
  Other Names: tiotropium: Spiriva
  Arms: 2

SUMMARY:
Study title

* A randomized, open label, multicenter, phase 4 study for the comparison of efficacy of tiotropium plus salmeterol/ fluticasone propionate compared with tiotropium alone in COPD patients

Study objectives

* To investigate clinical outcomes of combining tiotropium with fluticasone propionate/salmeterol (FSC) 250/50μg bid compared with tiotropium alone in patients with moderate or severe COPD in Korea

Study Design

* Randomized, open-label, multicenter, parallel-group, two group study

Study assessment

* FEV1
* Inspiratory capacity (IC)
* History of COPD exacerbation
* History of hospitalization for COPD exacerbation and all causes
* QoL (SGRQ-C)

ELIGIBILITY:
Inclusion Criteria:

* Subjects Aged 40 to 80 years.
* Subjects diagnosed with COPD.
* Tobacco smoking 10 pack-years or more.
* Subjects with post-bronchodilator FEV1/FVC < 0.7 and FEV1 < 65% predicted.

Exclusion Criteria:

* Subjects with a history of physician-diagnosed asthma or a respiratory disorder other than COPD which is clinically significant such as diffuse bilateral bronchiectasis.
* Subjects suffering from serious diseases likely to interfere with the study such as chronic congestive heart failure.
* Subjects who used systemic corticosteroids within 4 weeks prior to study entry.
* Subjects with any malignant disease.
* Subjects with a history of severe glaucoma, urinary tract obstruction.
* Previous lung volume reduction surgery.
* Subjects who are pregnant or breastfeeding.
* Subjects with a known hypersensitivity or intolerance to tiotropium or fluticasone-salmeterol.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 509 (Actual)
Dates: Start 2009-03; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
Changes in pre-dose FEV1 from baseline at 24 weeks after treatment | 24 weeks

SECONDARY OUTCOMES:
Changes in pre-dose FEV1 from baseline and IC from baseline, COPD exacerbation, QoL and safety | 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Jee-Hong Yoo, Professor, Principal Investigator — East West Neo Medical Center; Sang-Do Lee, Professor, Principal Investigator — Asan Medical Center
Locations (32):
- South Korea (32):
  - Soonchunhyang University Bucheon Hospital, Bucheon-si
  - Inje university Pusan Paik hospital, Busan
  - Chonbuk national university hospital, Chunbuk
  - Keimyung university dongsan medical center, Daegu
  - Kyungpook national university hospital, Daegu
  - Yeungnam University Hospital, Daegu
  - Hallym University scared heart hospital, Gyeonggi-do
  - Gachon University Gil Hospital, Inchon
  - Incheon St. Mary's Hospital, Inchon
  - Inha university Hospital, Inchon
  - Gyeongsang national university hospital, Jinju
  - Chungbuk national university hospital, Jungbuk
  - Chungnam National University Hospital, Jungnam
  - Kyunghee university east-west neo medical center, Seoul
  - Asan Medical Center, Seoul
  - Boramae Medical Center, Seoul
  - Ewha womans university mokdong hospital, Seoul
  - Hanyang University Hospital, Seoul
  - Inje university Seoul Paik Hospital, Seoul
  - Kangdong Scared heart Hospital, Seoul
  - Kangnam St. Mary's Hospital, Seoul
  - Konkuk university hospital, Seoul
  - Korea University Guro Hospital, Seoul
  - Kyunghee university medical center, Seoul
  - Samsung medical center, Seoul
  - Seoul National University Hospital, Seoul
  - Severance Hospital, Seoul
  - Soonchunhyang University hospital, Seoul
  - St. Paul's Hospital, Seoul
  - Ajou university hospital, Suwon
  - Uijeongbu St. Mary's Hospital, Uijeongbu-si
  - Wonju Christian Hospital, Wŏnju